CLINICAL TRIAL: NCT04505852
Title: Implementing Artificial-intelligence Wristbands to Help in Recording Seizures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, PEIYUAN F. HSIEH, Principal Investigator, Taichung Veterans General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CF19347A
Record Dates: First submitted 2020-08-05; First posted 2020-08-10 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EMBRACE USERS (Experimental): Embrace wristband users
  Interventions: Device: Embrace

INTERVENTIONS:
Device: Embrace — Patients wear Embrace2 to help in seizure reporting and patient care.

SUMMARY:
The investigators hypothesize that the participants will be satisfied with artificial-intelligence wristband Embrace

DETAILED DESCRIPTION:
Currently, seizure tracking relies on subjective patient and family recall. In several studies patients report only approximately half of their seizures, and even less during sleep.

Sudden unexplained death in epilepsy (SUDEP) is the cause of premature death of up to 17% of all patients with epilepsy and as many as 50% with chronic refractory epilepsy (with rates as high as 1% per year). Its etiology is probably due to peri-ictal respiratory, cardiac, or autonomic nervous system dysfunction.

Wristband sensors help caregivers assist patients during seizures and may reduce risks for complications such as injuries and SUDEP.

Accurate seizure detection may improve the quality of life (QoL) of subjects and caregivers by decreasing burden of seizure monitoring and may facilitate diagnostic monitoring in the home setting. Possible risks are occurrence of alarm fatigue and invasion of privacy.

The wristband Embrace has an overall sensitivity of 89.1% and an overall specificity of 93.1%. The investigators hypothesize that the participants will be satisfied with artificial-intelligence wristband Embrace.

Methods:

When the smart wristband detects the seizure, the mobile phone sends a text message to the companion and the nurse, the latter will see or get in touch with the companion and keep a record.

In-patients receiving video-electroencephalography (VEEG) exam use Embrace during the VEEG recording which usually takes 3-5 days.

Out-patients use Embrace for 8 weeks. The investigators will enroll 30-50 patients, half in-patients and half out-patients.

The benefits are evaluated in terms of satisfaction. .

ELIGIBILITY:
Inclusion Criteria:

* At least one seizure per month in the 3-month period before entering the study

Exclusion Criteria:

* Uncountable seizures, psychogenic seizures, alcohol or drug abuse, severe heart or lung disorder, rapid progressive brain disorder, life-terminal disease, severe infection/ bleeding/ liver/ kidney disorder, platelet <80,000/μL, neutrophil <1,000/μL, clinically significant ECG abnormality, unstable psychiatric disease (except anxiety).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Satisfaction score of seizure wristband | Through study completion, an average of 1 year
  Scores 1(least satisfied) to 10 (most satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: PEIYUAN F. HSIEH, MD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No